CLINICAL TRIAL: NCT05356676
Title: Effects of Progressive Cervical Isometric Exercises Versus Scapular Stabilization Exercises on Pain, Range of Motion and Disability in Young Adults With Text Neck Syndrome: A Randomised Controlled Trail
Brief Title: Progressive Cervical Isometric Exercises Versus Scapular Stabilization Exercises in Text Neck Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0112 Osama
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Neck Syndrome
Keywords: progressive cervical neck isometrics; scapular stabilization exercises; pain; ROM; Text neck syndrome; turtle neck syndrome; disability
MeSH Terms: conditions — Pain | interventions — Exercise; Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometrics (Experimental): They will be treated with progressive isometric exercises added to 60 min of combined therapy (excluding scapular stabilizing exercises) treatment session at alternative 3 days/week for 8weeks
  Interventions: Other: Isometrics
- Combination Therapy (Experimental): They will be treated with both isometric and scapular stabilizing exercises.and will get 60minutes of treatment sessions at alternative 3 days/week for 8weeks
  Interventions: Other: Combination Therapy

INTERVENTIONS:
Other: Isometrics — Isometric neck extension -individuals will be taught to place their dominant hand posterior to their head at occiput. Then, they will be told to firmly push the head backwards against that hand, and hold for five seconds and repeat 5 times. • Participants will be asked to place the right hand flat on the same side of the head. Next.
  they will be instructed to firmly push the head against right hand and hold for 5 seconds and repeat five times. Same exercise will be repeated with the left hand against the left side of the head as well.
  • Participants will be taught to place their right hand on their right cheek. Then, they will be told to rum the face against the right hand and wait for 5 seconds and repeat five times. Same exercise was repeated with the left hand on the left cheek as well.
  Arms: Isometrics
Other: Combination Therapy — 1. In supine position, the patient will be instructed to take a deep breath in order to relax the body whilst holding his/her shoulders and neck in a comfortable posture.
  2. the patient will bend his/her knees and place their feet flat on the floor, and will hold the posture without any other neck movement. Then the patient will be asked to raise their dominant arm to 90° shoulder flexion along with full elbow extension and scapular protraction.
     This posture will be held for 10 seconds before returning to the prior position with 3 laps, 10 repetitions with a one-minute break between.
  3. in quadruped position, the patient will lift up their arms alternatively with shoulder abduction and 120 ° flexion. This posture will be held for 10 seconds before returning to the starting position for three laps, 10 repetitions with a 30-second break in between. Participants will be instructed to perform these for 3 times a week for 4 weeks.
  Arms: Combination Therapy

SUMMARY:
The aim of this study is to investigate the effects of progressive cervical isometric exercises and scapular stabilization exercises on pain, ROM and disability in young adults with text neck syndrome.

DETAILED DESCRIPTION:
Text neck or Turtle neck posture is the latest term coined by Dr. Dean L. Fishman that demonstrates the repeated stress, injury, and pain in the neck due to having the head in a forward position by excessive use of cell phones or hand-held mobile devices for a prolonged time. The use of mobile devices is becoming a concern especially in children, recent numbers are very alarming and according to surveys 87% of teenagers in America and 79% of teenagers in the UK are mobile phone owners and are greatly affected by them, these numbers have skyrocketed by recent COVID-19 pandemic as the social distancing and closure of the school, colleges and offices have pushed us to work from home and it increases the prevalence of text neck syndrome. This study is unique in that as it investigate the effect of two different treatment plans for turtle neck syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Individuals using mobile phones for more than 6-8 hours.

  * Participants both male and female of age between 18 to 28 years
  * Participants with neck pain (>7 weeks)
  * Participants with NDI score above 15/50 (10% or higher) or
  * Participants with NPRS score above 3

Exclusion Criteria:

* Specific causes of neck pain (conditions with neurological involvement such as myelopathy with weakness, numbness and sensory loss, cervical disc prolapse, and cervical spinal stenosis)

  * Previous neck and upper limb surgery.
  * History of cervical trauma (whiplash disorder), fractures, dislocations.
  * History of congenital torticollis, frequent migraine, carcinoma, acute pain and inflammation, torticollis, unstable/acute osteoarthritis, any recent fracture, vertigo, vertebrobasilar insufficiency, chronic heart disease, myocardial infarction or pregnancy

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
NDI (Neck disability Index) | 3 months
  The Neck Disability Index (NDI) is modification of the Oswestry Low Back Pain Disability Index. It is Patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation
NPRS (Numeric Pain Rating Scale) | 3 months
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. Similar to the VAS, the NPRS is anchored by terms describing pain severity extremes
Goniometer | 3 months
  A goniometer is an instrument that either measures an angle or allows an object to be rotated to a precise angular position
Inclinometer | 3 months
  An inclinometer is a medical device used to measure the range of motion of the joint. They are mainly used to measure the passive range of motion and allow the medical practitioner to compare the patient's relaxed position to the ability to move

CONTACTS AND LOCATIONS:
Overall Officials: Nosheen Manzoor, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Services hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No